CLINICAL TRIAL: NCT04628325
Title: Effects of Treatment With Intravenous Furosemide Plus Small Hypertonic Saline Solutions (HSS) on Atrial Stretching, Fibrosis and Inflammatory Markers in Subjects With Heart Failure With Reduced Ejection Fraction.
Brief Title: Effects of Furosemide Plus Small HSS in Subjects With Heart Failure With Reduced Ejection Fraction (HFrEF)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Antonino Tuttolomondo, Professor, University of Palermo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UPalermo
Record Dates: First submitted 2020-11-02; First posted 2020-11-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Heart Failure，Congestive
Keywords: Congestive Heart Failure; HFrEF; Biomarkers; Inflammation; Atrial Stretching; Furosemide
MeSH Terms: conditions — Heart Failure; Inflammation | interventions — Furosemide

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high dose furosemide plus HSS (Experimental): Patients treated high dose furosemide plus HSS
  Interventions: Drug: Furosemide
- high dose furosemide alone (Active Comparator): Patients treated high dose furosemide alone
  Interventions: Drug: Furosemide

INTERVENTIONS:
Drug: Furosemide — Intravenous Furosemide Plus Small Hypertonic Saline Solutions (HSS)
  Other Names: Furosemide plus HSS

SUMMARY:
The investigators sought to evaluate the effectiveness of treatment with furosemide + HSS in terms of reduction of serum levels of some chosen markers of heart failure and the response in terms of these markers at a compensated state after an acute saline load.

DETAILED DESCRIPTION:
All consecutive patients aged >18 years with a diagnosis of acute heart failure or exacerbation in chronic heart failure due to heart failure with reduced ejection fraction ( HFrEF) admitted to the ward of Internal Medicine were enrolled from March 2017 to June 2019. Enrolled subjects were treated with treatment with hypertonic saline solutions + furosemide e.v and control subjects with congestive heart failure randomized to treatment with intravenous furosemide only. Chronic kidney disease patients undergoing dialysis replacement, acute coronary syndrome, myocarditis, pneumonia, myopathies, neoplasms have been excluded.

Patients underwent at T0 (at 24 hours from admission), T1 (after 6-8 days after treatment with high dose furosemide+ HSS ), T2 (after a saline load) venepuncture to obtain venous blood samples for the determination of serum concentrations of N terminal pro B-type natriuretic peptide, High-sensitive cardiac troponin T, Galectin 3, IL-6.

ELIGIBILITY:
Inclusion Criteria:

* Congestive Heart Failure

Exclusion Criteria:

* Acute myocarditis
* active pulmonary or liver diseases
* autoimmune disorders
* infections
* malignant diseases
* muscle disorders
* renal insufficiency
* chronic inflammatory diseases
* rheumatological diseases
* haematological diseases
* chronic treatment with anti-inflammatory drugs

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2020-05-01 (Actual)

PRIMARY OUTCOMES:
Effects of Treatment With Moderate/High Doses of Intravenous Furosemide Plus Small Hypertonic Saline Solutions (HSS) on Atrial Stretching | 6 days
  Assessment of differences between participants on atrial diameters evaluated with echocardiography
Effects of Treatment With Moderate/High Doses of Intravenous Furosemide Plus Small Hypertonic Saline Solutions (HSS) on Atrial Fibrosis | 6 days
  Assessment of differences between participants on atrial fibrosis evaluated with echocardiography
Effects of Treatment With Moderate/High Doses of Intravenous Furosemide Plus Small Hypertonic Saline Solutions (HSS) on Inflammatory Markers | 6 days
  Evaluation of serum level of cytokines linked to inflammation and cardiac damage (IL-6, High-sensitive cardiac troponin T, Soluble interleukin 1 receptor-like 1, Galectin-3, N Terminal proB-type natriuretic peptide, C Reactive Protein)

CONTACTS AND LOCATIONS:
Overall Officials: Antonino Tuttolomondo, PhD, Study Director — Internal Medicine and Stroke Care Ward, University of Palermo, Italy
Locations (2):
- Italy (2):
  - AOUP Paolo Giaccone, Palermo
  - Internal Medicine Ward of Palermo University Hospital, Palermo